CLINICAL TRIAL: NCT07027254
Title: A Randomized Controlled Trial to Evaluate the Effect of Gallium-68 Pentixafor PET-CT on Surgical Outcomes in Patients With Primary Aldosteronism (The PETAL Trial)
Brief Title: PETAL Trial: Impact of Gallium-68 Pentixafor PET-CT on Surgical Outcomes in Primary Aldosteronism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Su-jin Kim, Professor, Department of Surgery, Seoul National University Hospital, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2502-040-1612
Record Dates: First submitted 2025-06-04; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Primary Aldosteronism; Secondary Hypertension; Aldosterone-Producing Adenoma; Idiopathic Hyperaldosteronism; Adrenalectomy
Keywords: Primary aldosteronism; Gallium-68 pentixafor; 11C-metomidate; PET/CT; adrenal venous sampling; PASO; PAMO; Adrenalectomy
MeSH Terms: conditions — Hyperaldosteronism; Adrenocortical Adenoma

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The nuclear medicine physician interpreting PET/CT scans is masked to AVS results. However, participants and treating clinicians are not blinded due to the nature of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AVS + 68Ga-pentixafor PET/CT (+ 11C-metomidate PET/CT) (Experimental): Intervention:
  Diagnostic Imaging: 68Ga-pentixafor PET/CT
  With 68Ga-pentixafor PET/CT imaging added to AVS for lateralization Subset only: 11C-metomidate PET/CT (for research use only, not used in treatment decisions)
  Interventions: Diagnostic Test: 68Ga-pentixafor PET/CT
- AVS only (No Intervention): No PET/CT Without 68Ga-pentixafor PET/CT imaging; AVS only (Gold standard)

INTERVENTIONS:
Diagnostic Test: 68Ga-pentixafor PET/CT — Diagnostic PET/CT imaging using gallium-68 labeled pentixafor to assess adrenal CXCR4 expression in patients with primary aldosteronism. The imaging is performed prior to treatment allocation and used to assist lateralization of aldosterone production when combined with adrenal venous sampling (AVS).
  Arms: AVS + 68Ga-pentixafor PET/CT (+ 11C-metomidate PET/CT)

SUMMARY:
This study is a randomized controlled trial to assess the clinical utility of gallium-68 pentixafor PET/CT in the management of primary aldosteronism (PA). We aim to evaluate whether the addition of 68Ga-pentixafor PET/CT to standard adrenal venous sampling (AVS) improves surgical outcomes in patients with unilateral PA.

DETAILED DESCRIPTION:
Primary aldosteronism (PA) is a common cause of secondary hypertension. Accurate subtype classification (unilateral vs. bilateral) is essential to determine whether patients should receive adrenalectomy or medical therapy. AVS is the current gold standard but has limitations, including its invasiveness, technical difficulty, and risk of failure. Recently, non-invasive imaging techniques such as 68Ga-pentixafor PET/CT and 11C-metomidate PET/CT have emerged as promising alternatives for subtype classification. These PET-based methods target molecular markers (e.g., CXCR4, CYP11B2) and show moderate to high concordance rates with AVS (66.7%-90% for pentixafor). However, there is insufficient prospective evidence on whether these modalities can improve treatment outcomes. This randomized controlled trial aims to assess whether adding 68Ga-pentixafor PET/CT to standard AVS improves surgical outcomes in patients with unilateral PA. Participants are randomized 1:1 to undergo either AVS alone or AVS plus 68Ga-pentixafor PET/CT. Additionally, 11C-metomidate PET/CT is performed in the intervention arm purely for research purposes and will not influence treatment decisions. By improving the precision of subtype classification, this study aims to improve patient selection for adrenalectomy, and ultimately enhance clinical outcomes in primary aldosteronism.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥19 years
* Diagnosed with PA per 2016 Endocrine Society guidelines
* Underwent adrenal CT
* Signed informed consent

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or may become pregnant
* Individuals who refuse to undergo surgery
* Individuals for whom 68Ga-Pentixafor PET/CT, 11C-Metomidate PET/CT, or adrenal venous sampling (AVS) is not feasible or is refused due to underlying conditions
* Individuals who refuse or experience adverse effects from dexamethasone premedication required for 11C-Metomidate PET/CT
* Individuals with a history of abdominal open surgery or retroperitoneal surgery on the same side as the planned adrenalectomy
* Any individual deemed unsuitable for the study at the discretion of the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Biochemical remission rate after adrenalectomy (surgery group only) | 6 months after adrenalectomy
  Number of participants achieving biochemical success as defined by PASO criteria will be assessed. Biochemical success is defined as normalization or improvement in aldosterone-to-renin ratio (ARR) and correction of hypokalemia without potassium supplementation in patients with unilateral primary aldosteronism who underwent adrenalectomy.

SECONDARY OUTCOMES:
Clinical remission rate after adrenalectomy or initiation of medical therapy | 6 months after treatment (surgery or medication)
  Number of participants achieving clinical success according to PASO (surgical group) or PAMO (medical group) criteria will be assessed. Clinical success includes normalization of blood pressure and reduction in number or dose of antihypertensive medications after surgery or medical therapy.
Agreement rate between PET/CT imaging and adrenal venous sampling (AVS) | 6 months after treatment (surgery or medication)
  Agreement rate between 68Ga-pentixafor PET/CT (+11C-metomidate PET/CT for subgroup) and adrenal venous sampling (AVS) will be assessed. Diagnostic agreement will be evaluated based on lateralization patterns from PET/CT and AVS using predefined laterality thresholds.
Concordance between AVS-based lateralization and immunohistochemical (IHC) expression of CXCR4 and CYP11B2 | 6 months after treatment
  Concordance between AVS-based lateralization and immunohistochemical (IHC) expression of CXCR4 and CYP11B2 will be assessed. IHC positivity for CXCR4 and CYP11B2 will be recorded as presence or absence in each adrenal lesion. Concordance will be evaluated by comparing lateralization results from AVS with the presence or absence of expression.
Concordance between PET/CT-based lateralization and immunohistochemical (IHC) expression of CXCR4 and CYP11B2 | 6 months after treatment
  Concordance between PET/CT-based lateralization and immunohistochemical (IHC) expression of CXCR4 and CYP11B2 will be assessed. IHC positivity for CXCR4 and CYP11B2 will be recorded as presence or absence in each adrenal lesion. Concordance will be evaluated by comparing PET/CT-based lateralization with the presence or absence of expression in the corresponding adrenal tissue.
Correlation between the AVS-derived lateralization index and the SUVmax ratio on PET/CT | 6 months after treatment
  The correlation between the AVS-derived lateralization index and the SUVmax ratio on PET/CT will be evaluated. SUVmax ratios will be quantitatively compared with AVS findings, including the lateralization index, as well as tumor size and the side of dominant hormone secretion
Change in plasma aldosterone concentration/aldosterone-to-renin ratio (ARR) | Baseline and 6 months after treatment
  Change from baseline in plasma aldosterone concentration and ARR will be assessed. Plasma aldosterone and ARR will be measured at baseline and 6 months post-treatment to evaluate endocrine improvement.
Rate of blood pressure normalization | 6 months after treatment
  Proportion of participants with blood pressure below 140/90 mmHg without escalation of antihypertensive medications will be assessed. Participants achieving target blood pressure without medication escalation will be recorded.
Change in antihypertensive medication use | Baseline and 6 months after treatment
  Change in number and dose of antihypertensive medications from baseline will be assessed. Total daily defined dose and number of medications will be compared between baseline and 6 months after treatment.
Change in serum potassium level | Baseline and 6 months after treatment
  Change in serum potassium concentration from baseline will be assessed. Serum potassium levels at baseline and 6 months post-treatment will be compared to evaluate metabolic improvement.
Frequency and percentage of histologic subtype classification in resected adrenal tissue | 3 months after adrenalectomy
  Frequency and percentage of histologic subtype classification in resected adrenal tissue will be assessed. Resected adrenal tissues will be classified according to histologic subtypes, and the distribution of each subtype will be recorded.
Size of resected adrenal tumors | 3 months after adrenalectomy
  Size of resected adrenal tumors will be assessed. Tumor diameter will be measured in centimeters based on pathology reports.
Correlation between somatic mutations and PET/CT SUVmax ratio | 3 months after adrenalecotmy
  The correlation between somatic mutations and PET/CT SUVmax ratios of adrenal tumors will be evaluated. Mutation profiles (e.g., KCNJ5, CACNA1D, etc.) will be analyzed in relation to SUVmax measurements obtained from PET/CT imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Su-jin Kim, M.D, Ph.D, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Samsung Medical Center, Seoul, Gangnam-gu
  - Seoul National University Hospital, Seoul, Jongno-gu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim JH, Ahn CH, Kim SJ, Lee KE, Kim JW, Yoon HK, Lee YM, Sung TY, Kim SW, Shin CS, Koh JM, Lee SH. Outcome-Based Decision-Making Algorithm for Treating Patients with Primary Aldosteronism. Endocrinol Metab (Seoul). 2022 Apr;37(2):369-382. doi: 10.3803/EnM.2022.1391. Epub 2022 Apr 14. PMID 35417953
- [Background] Ren X, Cheng G, Wang Z. Advances in the molecular imaging of primary aldosteronism. Ann Nucl Med. 2023 Aug;37(8):433-441. doi: 10.1007/s12149-023-01851-y. Epub 2023 Jul 2. PMID 37393373
- [Background] Soinio M, Luukkonen AK, Seppanen M, Kemppainen J, Seppanen J, Pienimaki JP, Leijon H, Vesterinen T, Arola J, Lantto E, Helin S, Tikkanen I, Metso S, Mirtti T, Heiskanen I, Norvio L, Tiikkainen M, Tikkanen T, Sane T, Valimaki M, Gomez-Sanchez CE, Porsti I, Nuutila P, Nevalainen PI, Matikainen N. Functional imaging with 11C-metomidate PET for subtype diagnosis in primary aldosteronism. Eur J Endocrinol. 2020 Dec;183(6):539-550. doi: 10.1530/EJE-20-0532. PMID 33055298
- [Background] Burton TJ, Mackenzie IS, Balan K, Koo B, Bird N, Soloviev DV, Azizan EA, Aigbirhio F, Gurnell M, Brown MJ. Evaluation of the sensitivity and specificity of (11)C-metomidate positron emission tomography (PET)-CT for lateralizing aldosterone secretion by Conn's adenomas. J Clin Endocrinol Metab. 2012 Jan;97(1):100-9. doi: 10.1210/jc.2011-1537. Epub 2011 Nov 23. PMID 22112805
- [Background] Heinze B, Fuss CT, Mulatero P, Beuschlein F, Reincke M, Mustafa M, Schirbel A, Deutschbein T, Williams TA, Rhayem Y, Quinkler M, Rayes N, Monticone S, Wild V, Gomez-Sanchez CE, Reis AC, Petersenn S, Wester HJ, Kropf S, Fassnacht M, Lang K, Herrmann K, Buck AK, Bluemel C, Hahner S. Targeting CXCR4 (CXC Chemokine Receptor Type 4) for Molecular Imaging of Aldosterone-Producing Adenoma. Hypertension. 2018 Feb;71(2):317-325. doi: 10.1161/HYPERTENSIONAHA.117.09975. Epub 2017 Dec 26. PMID 29279316
- [Background] Umakoshi H, Naruse M, Wada N, Ichijo T, Kamemura K, Matsuda Y, Fujii Y, Kai T, Fukuoka T, Sakamoto R, Ogo A, Suzuki T, Nanba K, Tsuiki M; WAVES-J Study Group. Adrenal Venous Sampling in Patients With Positive Screening but Negative Confirmatory Testing for Primary Aldosteronism. Hypertension. 2016 May;67(5):1014-9. doi: 10.1161/HYPERTENSIONAHA.115.06607. Epub 2016 Mar 14. PMID 26975712
- [Background] Rossi GP, Auchus RJ, Brown M, Lenders JW, Naruse M, Plouin PF, Satoh F, Young WF Jr. An expert consensus statement on use of adrenal vein sampling for the subtyping of primary aldosteronism. Hypertension. 2014 Jan;63(1):151-60. doi: 10.1161/HYPERTENSIONAHA.113.02097. Epub 2013 Nov 11. PMID 24218436
- [Background] Hannemann A, Wallaschofski H. Prevalence of primary aldosteronism in patient's cohorts and in population-based studies--a review of the current literature. Horm Metab Res. 2012 Mar;44(3):157-62. doi: 10.1055/s-0031-1295438. Epub 2011 Dec 1. PMID 22135219
- [Background] Rossi GP, Bernini G, Caliumi C, Desideri G, Fabris B, Ferri C, Ganzaroli C, Giacchetti G, Letizia C, Maccario M, Mallamaci F, Mannelli M, Mattarello MJ, Moretti A, Palumbo G, Parenti G, Porteri E, Semplicini A, Rizzoni D, Rossi E, Boscaro M, Pessina AC, Mantero F; PAPY Study Investigators. A prospective study of the prevalence of primary aldosteronism in 1,125 hypertensive patients. J Am Coll Cardiol. 2006 Dec 5;48(11):2293-300. doi: 10.1016/j.jacc.2006.07.059. Epub 2006 Nov 13. PMID 17161262
- [Background] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393